CLINICAL TRIAL: NCT03278873
Title: Long-term Follow-up Study of Participants Following an Open Label, Multi-centre, Phase I/II Dose Escalation Trial of a Recombinant Adeno-associated Virus Vector (AAV2/8-hCARp.hCNGB3 and AAV2/8-hG1.7p.coCNGA3) for Gene Therapy of Adults and Children With Achromatopsia Owing to Defects in CNGB3 or CNGA3
Brief Title: Long-Term Follow-Up Gene Therapy Study for Achromatopsia CNGB3 and CNGA3
Status: Terminated | Type: Observational
Why Stopped: Strategic decision to not further develop AAV8-hCARp.hCNGB3 and AAV8-hG1.7p.coCNGA3. The decision is not due to safety concerns.
Sponsor: MeiraGTx UK II Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: MGT007; 2016-003856-59 (EudraCT Number)
Record Dates: First submitted 2017-08-16; First posted 2017-09-12 (Actual); Results first posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Achromatopsia
Keywords: Achromatopsia; CNGA3; CNGB3
MeSH Terms: conditions — Color Vision Defects

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Low dose of AAV-CNGA3 or AAV-CNGB3: Subretinal administration of a single low dose of AAV-CNGA3 or AAV-CNGB3
  Interventions: Biological: Prior exposure to AAV-CNGA3 or AAV-CNGB3
- Intermediate dose of AAV-CNGA3 or AAV-CNGB3: Subretinal administration of a single intermediate dose of AAV-CNGA3 or AAV-CNGB3
  Interventions: Biological: Prior exposure to AAV-CNGA3 or AAV-CNGB3
- Other dose of AAV-CNGA3 or AAV-CNGB3: Subretinal administration of a single other dose (between the intermediate and high dose) of AAV-CNGA3 or AAV-CNGB3
  Interventions: Biological: Prior exposure to AAV-CNGA3 or AAV-CNGB3
- High dose of AAV-CNGA3 or AAV-CNGB3: Subretinal administration of a single high dose of AAV-CNGA3 or AAV-CNGB3
  Interventions: Biological: Prior exposure to AAV-CNGA3 or AAV-CNGB3

INTERVENTIONS:
Biological: Prior exposure to AAV-CNGA3 or AAV-CNGB3 — Participants previously received AAV-CNGA3 or AAV-CNGB3 in an open-label, Phase 1/2 dose escalation trial for adults and children with achromatopsia owing to defects in CNGA3 or CNGB3, respectively.

SUMMARY:
This is a longer-term follow-up study of patients with achromatopsia associated with defects in CNGA3 who participated in a clinical trial in which they received AAV-CNGA3 retinal gene therapy, or of patients with achromatopsia associated with defects in CNGB3 who participated in a clinical trial in which they received AAV-CNGB3 retinal gene therapy.

DETAILED DESCRIPTION:
The follow-up study is designed to collect data on the longer-term safety and efficacy of AAV-CNGA3 retinal gene therapy and AAV-CNGB3 retinal gene therapy.

ELIGIBILITY:
Inclusion in the study will be limited to individuals who:

1. Are able to give informed consent or assent, with or without the guidance of their parent(s)/guardian(s), where appropriate
2. Received AAV2/8-hCARp.hCNGB3 or AAV2/8-hG1.7p.coCNGA3 by intraocular administration in the prior open-label, Phase I/II, dose escalation study (EudraCT 2016-002290-35 or EudraCT 2018-003431-29)
3. Are willing to adhere to the protocol and long-term follow-up

Individuals will be excluded who:

Are unwilling or unable to meet the requirements of the study

Ages: 3 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population are adults and children with achromatopsia resulting from mutations in CNGA3 or CNGB3.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2024-04-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Kellogg Eye Center, Ann Arbor, Michigan, United States
- Moorfields Eye Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from medical centers in the United Kingdom (UK) and the United States (US). A total of 34 participants were enrolled in the study.
Groups:
- Low Dose of AAV-CNGA3 or AAV-CNGB3: Subretinal administration of a single low dose of adeno-associated virus AAV-CNGA3 or AAV-CNGB3
  AAV gene therapy for defects in the CNGA3 or CNGB3 gene, respectively.
- Intermediate Dose of AAV-CNGA3 or AAV-CNGB3: Subretinal administration of a single intermediate dose of adeno-associated virus AAV-CNGA3 or AAV-CNGB3
  AAV gene therapy for defects in the CNGA3 or CNGB3 gene, respectively.
- Other Dose of AAV-CNGA3 or AAV-CNGB3: Subretinal administration of a single other dose (between the intermediate and high dose) of adeno-associated virus AAV-CNGA3 or AAV-CNGB3
  AAV gene therapy for defects in the CNGA3 or CNGB3 gene, respectively.
- High Dose of AAV-CNGA3 or AAV-CNGB3: Subretinal administration of a single high dose of adeno-associated virus AAV-CNGA3 or AAV-CNGB3
  AAV gene therapy for defects in the CNGA3 or CNGB3 gene, respectively.
Period: Overall Study
Arm/Group | Low Dose of AAV-CNGA3 or AAV-CNGB3 | Intermediate Dose of AAV-CNGA3 or AAV-CNGB3 | Other Dose of AAV-CNGA3 or AAV-CNGB3 | High Dose of AAV-CNGA3 or AAV-CNGB3
Started | 6 | 15 | 3 | 10
Completed | 3 | 6 | 0 | 2
Not Completed | 3 | 9 | 3 | 8
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Sponsor's decision | 0 | 1 | 0 | 0
Not completed — Early Termination | 2 | 6 | 0 | 4
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0
Not completed — The patient decided to withdraw via email | 1 | 0 | 0 | 0
Not completed — The patient was unresponsive to contact | 0 | 0 | 0 | 4
Not completed — The patient wished to participate no longer | 0 | 1 | 0 | 0
Not completed — Patient withdrew as they could no longer participate, as they had moved to Canada | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Low Dose AAV-CNGA3 or AAV-CNGB3: Subretinal administration of a single low dose of adeno-associated virus AAV-CNGA3 or AAV-CNGB3
  AAV gene therapy for defects in the CNGA3 or CNGB3 gene, respectively.
- Intermediate Dose AAV-CNGA3 or AAV-CNGB3: Subretinal administration of a single intermediate dose of adeno-associated virus AAV-CNGA3 or AAV-CNGB3
  AAV gene therapy for defects in the CNGA3 or CNGB3 gene, respectively.
- Other Dose AAV-CNGA3 or AAV-CNGB3: Subretinal administration of a single other dose (between the intermediate and high dose) of adeno-associated virus AAV-CNGA3 or AAV-CNGB3
  AAV gene therapy for defects in the CNGA3 or CNGB3 gene, respectively.
- High Dose AAV-CNGA3 or AAV-CNGB3: Subretinal administration of a single high dose of adeno-associated virus AAV-CNGA3 or AAV-CNGB3
  AAV gene therapy for defects in the CNGA3 or CNGB3 gene, respectively.
- Total: Total of all reporting groups
Arm/Group | Low Dose AAV-CNGA3 or AAV-CNGB3 | Intermediate Dose AAV-CNGA3 or AAV-CNGB3 | Other Dose AAV-CNGA3 or AAV-CNGB3 | High Dose AAV-CNGA3 or AAV-CNGB3 | Total
Number analyzed (Participants) | 6 | 15 | 3 | 10 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 11 | 3 | 5 | 22
  Between 18 and 65 years | 3 | 4 | 0 | 5 | 12
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 10 | 3 | 4 | 20
  Male | 3 | 5 | 0 | 6 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 2 | 2
  Not Hispanic or Latino | 6 | 15 | 3 | 8 | 32
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 0 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 4 | 14 | 3 | 8 | 29
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 0 | 1 | 2 | 2 | 5
  United Kingdom | 6 | 14 | 1 | 8 | 29

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events Related to the Treatment
Description: The primary outcome measure is the longer-term safety of treatment with AAV-CNGA3 or AAV-CNGB3, assessed by the absence of IMP-related adverse events.
Time Frame: 5 Years
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose AAV-CNGA3 or AAV-CNGB3 | Intermediate Dose AAV-CNGA3 or AAV-CNGB3 | Other Dose AAV-CNGA3 or AAV-CNGB3 | High Dose AAV-CNGA3 or AAV-CNGB3
Number analyzed (Participants) | 6 | 15 | 3 | 10
Participants | 1 | 2 | 0 | 0

2. Secondary Outcome: Improvements in Visual Function as Assessed by Visual Acuity at Month 12
Description: Change from baseline to Month 12 in best corrected visual acuity (BCVA) using Early Treatment Diabetic Retinopathy Study (ETDRS) chart letter score in the treated eye. The direction of improvement from baseline is an increase in the number of ETDRS letters read over time.
Time Frame: 12 months
Population: 32 of the 34 participants performed the visual acuity assessment at baseline and Month 12.
Measure: Mean (Full Range); unit: Number of ETDRS letters
Arm/Group | Low Dose AAV-CNGA3 or AAV-CNGB3 | Intermediate Dose AAV-CNGA3 or AAV-CNGB3 | Other Dose AAV-CNGA3 or AAV-CNGB3 | High Dose AAV-CNGA3 or AAV-CNGB3
Number analyzed (Participants) | 6 | 15 | 2 | 9
Number of ETDRS letters | -0.6 [-3 to 1] | 0.2 [-5 to 4] | 3.5 [3 to 4] | 4.0 [-3 to 9]

3. Secondary Outcome: Improvements in Visual Function as Assessed by Visual Acuity at Month 60
Description: Change from baseline to Month 60 in best corrected visual acuity (BCVA) using Early Treatment Diabetic Retinopathy Study (ETDRS) chart letter score in the treated eye. The direction of improvement from baseline is an increase in the number of ETDRS letters read over time.
Time Frame: 60 months
Population: 16 of the 34 participants performed the visual acuity assessment at baseline and Month 60.
Measure: Mean (Full Range); unit: Number of ETDRS letters
Arm/Group | Low Dose AAV-CNGA3 or AAV-CNGB3 | Intermediate Dose AAV-CNGA3 or AAV-CNGB3 | Other Dose AAV-CNGA3 or AAV-CNGB3 | High Dose AAV-CNGA3 or AAV-CNGB3
Number analyzed (Participants) | 4 | 8 | 0 | 4
Number of ETDRS letters | 3.3 [-4 to 7] | 0.1 [-4 to 3] |  | -0.3 [-7 to 7]

4. Secondary Outcome: Improvements in Retinal Function as Assessed by Static Perimetry at Month 12
Description: Change from baseline to Month 12 in contrast sensitivity in the treated eye. The direction of improvement is an increase in sensitivity.
Time Frame: 12 months
Population: 31 of the 34 participants had contrast sensitivity data available at both baseline and Month 12 in the treated eye.
Measure: Mean (Full Range); unit: LogCS
Arm/Group | Low Dose AAV-CNGA3 or AAV-CNGB3 | Intermediate Dose AAV-CNGA3 or AAV-CNGB3 | Other Dose AAV-CNGA3 or AAV-CNGB3 | High Dose AAV-CNGA3 or AAV-CNGB3
Number analyzed (Participants) | 6 | 14 | 2 | 9
LogCS | -0.08 [-0.3 to 0.2] | -0.17 [-0.4 to 0.1] | 0.12 [0.0 to 0.2] | 0.03 [-0.2 to 0.3]

5. Secondary Outcome: Improvements in Retinal Function as Assessed by Static Perimetry at Month 60
Description: Change from baseline to Month 60 in contrast sensitivity in the treated eye. The direction of improvement is an increase in sensitivity.
Time Frame: 60 months
Population: 15 of the 34 participants had contrast sensitivity data available at both baseline and Month 60 in the treated eye.
Measure: Mean (Full Range); unit: LogCS
Arm/Group | Low Dose AAV-CNGA3 or AAV-CNGB3 | Intermediate Dose AAV-CNGA3 or AAV-CNGB3 | Other Dose AAV-CNGA3 or AAV-CNGB3 | High Dose AAV-CNGA3 or AAV-CNGB3
Number analyzed (Participants) | 4 | 7 | 0 | 4
LogCS | -0.19 [-1.0 to 0.4] | -0.11 [-0.4 to 0.1] |  | -0.12 [-0.3 to 0.1]

6. Secondary Outcome: Quality of Life at Month 12 Measured by QoL Questionnaires in Children and Adolescents
Description: Change from baseline to Month 12 in EuroQol-5D-Y Visual Analogue Scale (EQ-VAS) in children and adolescents. EQ-VAS uses a scale from 0 to 100, where 0 represents the worst imaginable health state and 100 represents the best imaginable health state. A positive change from baseline reflects improvement, and a negative change from baseline reflects worsening.
Time Frame: 12 months
Population: Eleven pediatric participants had EuroQol-5D-Y EQ-VAS data available at both baseline and Month 12. For this study outcome, pediatric participants are participants aged <16 years in the UK and aged <18 years in the US.
Measure: Mean (Full Range); unit: Units on a scale
Arm/Group | Low Dose AAV-CNGA3 or AAV-CNGB3 | Intermediate Dose AAV-CNGA3 or AAV-CNGB3 | Other Dose AAV-CNGA3 or AAV-CNGB3 | High Dose AAV-CNGA3 or AAV-CNGB3
Number analyzed (Participants) | 0 | 8 | 2 | 1
Units on a scale |  | 4.3 [-6 to 19] | 9.5 [9 to 10] | -12.0 [-12 to -12]

7. Secondary Outcome: Quality of Life at Month 60 Measured by QoL Questionnaires in Children and Adolescents
Description: Change from baseline to Month 60 in EuroQol-5D-Y Visual Analogue Scale (EQ-VAS) in children and adolescents. EQ-VAS uses a scale from 0 to 100, where 0 represents the worst imaginable health state and 100 represents the best imaginable health state. A positive change from baseline reflects improvement, and a negative change from baseline reflects worsening.
Time Frame: 60 months
Population: Two pediatric participants had EuroQol-5D-Y EQ-VAS data available at both baseline and Month 60. For this study outcome, pediatric participants are participants aged <16 years in the UK and aged <18 years in the US.
Measure: Mean (Full Range); unit: Units on a scale
Arm/Group | Low Dose AAV-CNGA3 or AAV-CNGB3 | Intermediate Dose AAV-CNGA3 or AAV-CNGB3 | Other Dose AAV-CNGA3 or AAV-CNGB3 | High Dose AAV-CNGA3 or AAV-CNGB3
Number analyzed (Participants) | 0 | 2 | 0 | 0
Units on a scale |  | 0.0 [-20 to 20] |  |

8. Secondary Outcome: Quality of Life at Month 12 Measured by QoL Questionnaires in Adults
Description: Change from baseline to Month 12 in EuroQol-5D-5L Visual Analogue Scale (EQ-VAS) in adults. EQ-VAS uses a scale from 0 to 100, where 0 represents the worst imaginable health state and 100 represents the best imaginable health state. A positive change from baseline reflects improvement, and a negative change from baseline reflects worsening.
Time Frame: 12 months
Population: Two adult participants had EuroQol-5D-5L EQ-VAS data available at both baseline and Month 12. For this study outcome, adults are participants aged ≥16 years in the UK and aged ≥18 years in the US.
Measure: Mean (Full Range); unit: Units on a scale
Arm/Group | Low Dose AAV-CNGA3 or AAV-CNGB3 | Intermediate Dose AAV-CNGA3 or AAV-CNGB3 | Other Dose AAV-CNGA3 or AAV-CNGB3 | High Dose AAV-CNGA3 or AAV-CNGB3
Number analyzed (Participants) | 0 | 0 | 0 | 2
Units on a scale |  |  |  | 0.5 [0 to 1]

9. Secondary Outcome: Quality of Life at Month 60 Measured by QoL Questionnaires in Adults
Description: Change from baseline to Month 60 in EuroQol-5D-5L Visual Analogue Scale (EQ-VAS) in adults. EQ-VAS uses a scale from 0 to 100, where 0 represents the worst imaginable health state and 100 represents the best imaginable health state. A positive change from baseline reflects improvement, and a negative change from baseline reflects worsening.
Time Frame: 60 months
Population: One adult participant had EuroQol-5D-5L EQ-VAS data available at both baseline and Month 60. For this study outcome, adults are participants aged ≥16 years in the UK and aged ≥18 years in the US.
Measure: Mean (Full Range); unit: Units on a scale
Arm/Group | Low Dose AAV-CNGA3 or AAV-CNGB3 | Intermediate Dose AAV-CNGA3 or AAV-CNGB3 | Other Dose AAV-CNGA3 or AAV-CNGB3 | High Dose AAV-CNGA3 or AAV-CNGB3
Number analyzed (Participants) | 1 | 0 | 0 | 0
Units on a scale | 0.0 [0 to 0] |  |  |

ADVERSE EVENTS:
Time Frame: 5 years
Groups:
- Total: Safety Analysis Set
Arm/Group | Low Dose AAV-CNGA3 or AAV-CNGB3 | Intermediate Dose AAV-CNGA3 or AAV-CNGB3 | Other Dose AAV-CNGA3 or AAV-CNGB3 | High Dose AAV-CNGA3 or AAV-CNGB3 | Total
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/15 | 0/3 | 0/10 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/15 | 0/3 | 1/10 | 2/34
Other Adverse Events (participants affected / at risk) | 1/6 | 4/15 | 3/3 | 2/10 | 10/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose AAV-CNGA3 or AAV-CNGB3 (N=6) | Intermediate Dose AAV-CNGA3 or AAV-CNGB3 (N=15) | Other Dose AAV-CNGA3 or AAV-CNGB3 (N=3) | High Dose AAV-CNGA3 or AAV-CNGB3 (N=10) | Total (N=34)
Retinal detachment (Eye disorders) | 0 | 1 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose AAV-CNGA3 or AAV-CNGB3 (N=6) | Intermediate Dose AAV-CNGA3 or AAV-CNGB3 (N=15) | Other Dose AAV-CNGA3 or AAV-CNGB3 (N=3) | High Dose AAV-CNGA3 or AAV-CNGB3 (N=10) | Total (N=34)
Vision blurred (Eye disorders) | 0 | 2 | 0 | 1 | 3
Dry eye (Eye disorders) | 0 | 2 | 0 | 0 | 2
influenza (Infections and infestations) | 0 | 1 | 2 | 0 | 3
COVID-19 (Infections and infestations) | 0 | 1 | 0 | 1 | 2
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1 | 0 | 2
Headache (Nervous system disorders) | 1 | 1 | 0 | 0 | 2

LIMITATIONS AND CAVEATS:
Upon agreement with the FDA, the study was prematurely terminated in March 2024. Therefore, the Month 60 data are not available for all participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-12-03): https://cdn.clinicaltrials.gov/large-docs/73/NCT03278873/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-22): https://cdn.clinicaltrials.gov/large-docs/73/NCT03278873/SAP_001.pdf